CLINICAL TRIAL: NCT07021053
Title: Adaptive Actions and Alcohol Use Outcomes During Internet-delivered Cognitive Behaviour Therapy: An Observational Study During Routine Care
Brief Title: Adaptive Actions and Alcohol Use Outcomes During Internet-delivered Cognitive Behaviour Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regina (Other)
Collaborators: Karolinska Institutet (Other); Macquarie University, Australia (Other); York University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-082b
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-05

CONDITIONS: Alcohol Misuse
Keywords: Internet-delivered cognitive behaviour therapy; Alcohol misuse
MeSH Terms: interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICBT for Alcohol Misuse (Experimental): Internet-delivered cognitive behavioral therapy for alcohol misuse.
  Interventions: Behavioral: Alcohol Change Course Enhanced

INTERVENTIONS:
Behavioral: Alcohol Change Course Enhanced — The Alcohol Change Course Enhanced is an adaptation of the Alcohol Change Course, originally developed and evaluated in Switzerland. The Course is a six-lesson ICBT intervention delivered over eight weeks to individuals who self-report alcohol misuse. Due to therapist registration and availability, eligible clients residing in Saskatchewan will be offered the option of receiving therapist assistance (or not) alongside the Course, while clients from other Canadian provinces will not receive therapist support. In addition to the monitoring of weekly measures available to all clients, those receiving therapist support will receive weekly secure messaging from their assigned therapist for eight weeks. Therapists will spend approximately 15 minutes per week/per client receiving therapist support. Phone calls will be used in the event that there is a significant clinical issue requiring therapist attention that cannot be addressed over messaging (e.g., sudden increase in symptoms).

SUMMARY:
This observational study investigates an Internet-delivered Cognitive Behaviour Therapy (ICBT) intervention for alcohol misuse, called the Alcohol Change Course Enhanced (ACCE). The intervention will be offered through the Online Therapy Unit, which is a routine care ICBT clinic. The primary objective of the study is to examine whether engagement in adaptive actions measured by the Things You Do Questionnaire (TYDQ), including healthy thinking, meaningful activities, social connections, healthy habits and goal setting - increase during ICBT for alcohol misuse. Using data collected during routine care, the relationship between adaptive actions and alcohol use will be investigated, and specifically explore if the frequency of adaptive actions increases as alcohol use reduces during the intervention.

DETAILED DESCRIPTION:
Internet-delivered Cognitive Behaviour Therapy (ICBT) is an effective intervention for a variety of psychological concerns, including alcohol misuse. In ICBT, clients access structured online content (e.g., lessons, worksheets), similar to the therapeutic content that is delivered in face-to-face cognitive behaviour therapy. ICBT can be offered with or without brief therapist support, which often involves the use of secure messaging. Past research shows that ICBT for alcohol misuse is effective both when self-guided and therapist-guided. Previous studies of an ICBT course for alcohol misuse (the Alcohol Change Course Enhanced) by the Online Therapy Unit found that clients report large reductions in weekly alcohol consumption and heavy drinking days. Further, clients report significant reductions in symptoms of anxiety and depression, cravings, risky or hazardous alcohol consumption, anger, PTSD, insomnia, and work and social adjustment.

An important body of work has demonstrated that individuals thoughts and daily actions have a significant impact on their psychological health. The Things You Do Questionnaire (TYDQ) was developed to capture the adaptive (i.e., helpful) actions most strongly associated with psychological health including: Healthy Thinking, Meaningful Activities, Goals and Plans, Healthy Habits, and Social Connections. Research shows that those who engage in the identified actions at least half of the days of the week report lower symptoms of depression and anxiety, and conversely, increased satisfaction with life. Subsequent research has shown that the frequency of these actions change during ICBT for depression and anxiety. Specifically, the frequency of adaptive actions increases across treatment, and increases in adaptive actions mirrors the decreases in depressive and anxiety symptoms over time.

For clients with alcohol misuse, the investigators assume that as these clients reduce alcohol use, they will also increase engagement in these behaviors that are known to be associated with psychological health, but this has not yet been systematically examined during ICBT. Engagement in adaptive actions may also help prevent relapse, such that if clients increase adaptive actions, they may be more likely to maintain reductions in alcohol use.

Of note, within the Online Therapy Unit, the ICBT for alcohol misuse program addresses TYD within the current treatment materials at various points. In the recent revision of the course, the investigators have highlighted how these actions are helpful for reducing alcohol use and are also associated with psychological health.

Lesson 1 - Provides alcohol psycho education and explains 5 Things You Do as helpful activities; highlights how Goal Setting is helpful for alcohol reduction and improving psychological health; Lesson 2 - Provides information on risk situations and seemingly unimportant decisions; highlights how Engaging in Meaningful Activities and Healthy Routines is helpful for alcohol reduction and improving psychological health; Lesson 3 - Discusses saying no and coping with cravings; highlights how Social Connection is helpful for alcohol reduction and improving psychological health; Lesson 4 - Discusses thought challenging; highlights how Healthy Thinking is helpful for alcohol reduction and improving psychological health; Lesson 5 - Discusses problem solving; highlights how Social Connection is helpful for alcohol reduction and improving psychological health; Lesson 6 - Discusses relapse prevention and planning for the future; highlights the importance of Goal Setting as helpful for alcohol reduction longer term and improving psychological health.

The primary aim of the current study will be to extend research on the TYD to ICBT for alcohol misuse. The investigators will explore the relationship between alcohol use and adaptive actions at pre-treatment and if the frequency of adaptive actions increases as alcohol problems improve. Observational data will be collected at pre-treatment, mid-treatment, post-treatment, and follow-up as part of routine care at the Online Therapy Unit, funded by the Saskatchewan government to provide ICBT to Saskatchewan residents. Saskatchewan clients who meet eligibility criteria will indicate their preference for the therapist-guided or self-guided (with monitoring) ACCE. Clients from other provinces in Canada will be offered self-guided ACCE only. Findings from this study may inform future enhancements to ICBT for alcohol misuse.

ELIGIBILITY:
Inclusion Criteria:

* Be a resident of Canada
* Be 18 years or older
* Have access to a computer or appropriate device and the internet
* Endorse alcohol misuse

Exclusion Criteria:

* Current severe medical or psychiatric problem that requires immediate or alternate treatment (e.g. current and recent mania or psychosis requiring hospitalization, actively suicidal and unable to keep themselves safe, medical condition requiring immediate surgery or other invasive treatment, severe substance use, severe cognitive impairment);
* Currently receiving or expecting to receive individual alcohol treatment more than twice per month
* Other treatment in our clinic
* Unable to read and understand English. (All content is provided in English and staff is English speaking; it is cost prohibitive at this time to provide the complete service in languages other than English)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2026-05-14 (Estimated); Study Completion 2026-05-14 (Estimated)

PRIMARY OUTCOMES:
Changes in Alcohol Consumption | Baseline (Screening), weeks 4, 6 (post-treatment) and 18 post enrollment
  Measured with Total Number of Drinks in the Last Week. Clients report the number of standard drinks consumed on each of the preceding 7 days, with numeric values. Two variables are derived for each time point (screening, mid-treatment, post-treatment, and follow-up): 1) total weekly consumption, calculated as the sum of standard drinks during the preceding 7 days, and 2) number of heavy drinking days (HDDs) in the past week. HDDs are defined as days on which consumption exceeds gender-specific thresholds defined by the National Institute on Alcohol Abuse and Alcoholism (i.e., 4 or more standard drinks for women, 5 or more for men).
Changes in Adaptive Actions | Baseline (Screening), weeks 4, 6 (post treatment) and 18 post enrollment
  Measured using the Things You Do Questionnaire-15 item (TYDQ-15), which consists of 15 items related to 5 factors: healthy thinking, meaningful activities, goals and plans, healthy habits, and social connections on a 5-point Likert scale ranging from 0-4. Scores are summed into subscale scores ranging from 0 to 12, and a total score ranging from 0 to 60, with higher scores indicating greater engagement in adaptive actions. Clients self-report how often they engaged in each activity in the last week.

SECONDARY OUTCOMES:
Changes in Alcohol Craving | Baseline(Screening), weeks 6 (post treatment) and 18 post enrollment
  Measured using the Penn Alcohol Cravings Scale. 5 items are measured on a 7-point Likert scale ranging from 0-6. Scores are summed into a total score ranging from 0 to 30. Higher scores indicate greater alcohol cravings.
Change in Alcohol Use Disorder Identification Test Scores | Baseline(Screening), weeks 6 (post-treatment) and 18 (follow up)
  The Alcohol Use Disorder Identification Test (AUDIT) is a10-item screening tool to assess for problematic alcohol use. The first eight items are measured on a 5-point Likert scale ranging from 0-4, while the last two items are measured on a 3-point Likert scale ranging from 0-4. 10 items are summed to produce a total score ranging from 0 to 40, with higher scores indicating more severe alcohol use problems.
Changes in Depression | Baseline (Screening), weeks 1, 4, 6 (post treatment) and 18 week post enrollment
  Measured using the Patient Health Questionnaire 9-item (PHQ-9). 9 items are measured on a 4-point Likert scale ranging from 0-3. Scores are summed for a total score ranging from 0 to 27. Higher scores indicate more severe depressive symptoms.
Changes in Anxiety | Baseline (Screening), weeks 6 and 18 post enrollment
  Measured using the Generalized Anxiety Disorder 7-item (GAD-7). 7 items are measured on a 4-point Likert scale ranging from 0-3. Scores are summed to create a total score ranging from 0 to 21, with higher scores indicating more severe symptoms.
Change in Anger | Baseline (Screening), weeks 6 and 18 post enrollment
  Measured using the Dimensions of Anger Reactions (DAR-5). 5 items are measured on a 5-point Likert scale ranging from 1-5. Scores are summed to produce a total score range from 5 to 25, with higher scores indicating greater severity of anger problems.
Changes in Loneliness | Baseline (Screening), weeks 6 and 18 post enrollment
  Measured using the UCLA 3-Item Loneliness Scale, which includes self-report items that measure three dimensions of loneliness (i.e., relational connectedness, social connectedness, and self-perceived isolation). 3 items are measured on a 3-point Likert scale ranging from 1-3. Scores are summed into a total score ranging from 3 to 9, with higher scores indicating greater feelings of loneliness.
Changes in Relationship Functioning | Baseline(Screening), weeks 6 and 18 post enrollment
  Measured using the Couples Satisfaction Index 4-item (CSI-4). The first item is measured on a 7-point Likert scale ranging from 0-6. The last three items are measured on a 6-point Likert scale ranging from 0-5. Scores are summed to produce a total score ranging from 0 to 21. Higher total scores indicate greater relationship satisfaction, with scores <13.5 indicating notable dissatisfaction.
Changes in Functioning | Baseline(Screening), weeks 6 and 18 week post enrollment
  Measured using the 5-item Work and Social Adjustment Scale (WSAS). 5 items are measured on a 9-point Likert scale ranging from 0-8. Scores are summed into a total score range from 0 to 40, with higher scores indicating more severe impairment in functioning. Scores of 10 or higher indicate moderate impairment. Scores of 20 or higher indicate severe impairment.
Changes in Treatment Credibility and Expectancy | Baseline (Screening), weeks 3 and 6 post treatment.
  Measured using the Credibility and Expectancy Questionnaire, which includes 6 items, with two subscales, to assess clients' beliefs about how credible and helpful a treatment will be for them. Each subscale contains 3-items. The three items of each subscale are measured on a 1-9 point Likert scale, with subscale scores ranging from 3 to 27. Higher scores in each sub-scale indicate greater treatment credibility or treatment expectancy respectively.
Structured Interview | Week 3
  Email invitation will be sent to clients (until saturation is met) during week 2 for them to schedule an appointment for a telephone interview with a member of the research team. Interviews will focus on collecting information about client expectancy and credibility of the course.

OTHER OUTCOMES:
Background Information | Baseline (Screening)
  Background information including demographic questions will be collected at screening for descriptive purposes. No scores are calculated.
Drug Use | Baseline(Screening)
  The Drug Use Disorder Identification Test-Concise (DUDIT-C) is a 4-item measure used to assess problematic drug use. Items are measured on a 5-point Likert scale ranging from 0-4, with total scores ranging from 0-16. Higher scores indicate more severe drug use problem.
Motivation for Change | Baseline (Screening)
  Measure of clients' motivation for changing their alcohol use. Clients self-report the importance of changing their alcohol use, their confidence in their ability to change their alcohol use, and their readiness to change their alcohol use using 3 items. Each item is rated from 1-10, and scores are summed to produce a total score ranging from 3-30, with higher scores indicating higher motivation.
Changes in Alcohol Consumption in the Previous Week | Weeks 1-3, 5, 7, 8
  Clients self-report how many total standard drinks they consumed in the previous week and the number of days they consumed alcohol using two questions. Standard drinks are defined as: one 12 oz (341 mL) can or bottle of 5% beer, cider, or cooler; one 4.5 oz (142 mL) glass of 12% wine; or one 1.3-1.5 oz (40-45 mL) shot of 40% distilled spirits. This measure is used by clinicians to assess alcohol consumption on weeks when the primary alcohol measures are not administered.
Alcohol Change Goal Questionnaire | Week 2 and 6 (post treatment)
  Measures clients' goals related to their alcohol use with two or three open-ended questions depending on whether client's goal is to quit or cut down alcohol consumption or some other goal. These questions explore what the maximum number of drinks will be if client's goal is to cut down alcohol consumption, other goals client have during the course, and what would help them in achieving their goals. This questionnaire was developed by the research team and does not have a sum score.
Homework Reflection | Weeks 2, 3, 4, 5, 6(post treatment), 7, 8
  A 5-item questionnaire assessing clients' week-to-week experiences in the ACCE, with items inquiring about the lesson participants worked on; effort exerted towards skills; helpfulness of lessons; and client successes, challenges and experiences over the previous week. A combination of checklist, Likert scale [7-point (1-7)], and open-ended response options are used to gauge participants' participation. This brief questionnaire has been developed by the research team and does not have a sum score.
Additional Resource Questions | Week 6(post-treatment)
  Clients are asked about their opinions of and satisfaction with the additional resources that they have reviewed since the beginning of the ACCE using yes/no dichotomous, multiple choice, and Likert scale response option. This questionnaire was developed by the research team and does not have a total score.
Evaluation of Treatment | Week 6 (post-treatment)
  A 12-item questionnaire used to assess satisfaction with treatment and negative effects experienced by clients during treatment. The questionnaire uses a combination of Likert-scale [5-point (0-4) and 6-point (0-5)], open-ended, and dichotomous yes/no response options to gauge participants' perceptions of the course. The questionnaire has been developed by the research team. A total score is not produced for this measure.
Other Forms of Help | Week 6 (post-treatment) and 18 post-enrollment
  Examines other types of help that clients received during treatment. This questionnaire has been developed by the research team and does not have a sum score.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Hadjistavropoulos, PhD, Principal Investigator — University of Regina
Locations (1):
- Online Therapy Unit, Regina, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No